CLINICAL TRIAL: NCT06849817
Title: PRO-WELL: Protein and Exercise for Postmenopausal Women's Wellbeing
Brief Title: Protein and Exercise for Postmenopausal Women's Wellbeing
Acronym: PROWELL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Associate Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PROWELL - 532739; AWD-104591 (Other: National Cattlemen's Beef Association)
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Postmenopausal
Keywords: Postmenopausal; Protein; Mood; Sleep; Wellbeing; Body composition; Amino acids
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Participants are free-living and are asked to follow their typical dietary pattern and physical activity pattern. Maintain protein consumption at 0.8 g protein /kg body weight or less and limit red meat consumption for 16 weeks.
- Protein (Beef) (Experimental): Participants will asked to consume beef 7 times per week (1 serving per day; 25 grams protein per serving (~100 grams beef) as part of a higher protein diet (1.6 g protein/kg body weight).
  Interventions: Other: Diet - higher protein
- Protein (Beef) + Physical Activity (Experimental): Participants will be asked to consume beef 7 times per week (1 serving per day; 25 grams protein per serving (~100 grams beef to yield 25 grams of protein)) as part of a higher protein diet (1.6 g protein/kg body weight) in combination with 150 minutes of physical activity including strength training 3 times per week.
  Interventions: Other: Diet - higher protein; Behavioral: Physical activity and resistance training

INTERVENTIONS:
Other: Diet - higher protein — Beef consumption 7 times per week (1 serving per day; 25 grams protein per serving (~100 grams beef) as part of a higher protein diet (1.6 g protein/kg body weight)
  Arms: Protein (Beef); Protein (Beef) + Physical Activity
Behavioral: Physical activity and resistance training — 150 minutes of physical activity including strength training 3 times per week
  Arms: Protein (Beef) + Physical Activity

SUMMARY:
The goal of this clinical trial is to learn if consuming a higher protein diet that includes one serving of beef each day, in combination with resistance exercise, improves wellbeing in postmenopausal women. It will also tell us about how higher protein intake changes body composition and blood values related to health. The main questions it aims to answer are:

* Does higher protein intake combined with resistance training improve mood and sleep in postmenopausal women?
* What other health benefits to postmenopausal women experience when the follow a higher protein diet and participate in resistance exercise?

Researchers will compare three groups 1) postmenopausal women living their daily lives as usual, 2) postmenopausal women consuming a higher protein diet, and 2) postmenopausal women consuming a higher protein diet and participating in resistance training.

Participants will:

* Consume a higher protein diet for 16 weeks
* Participate in an at-home resistance training for 16 weeks
* Keep a diary of their food intake, sleep habits, and mood
* Have health assessments every 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50 years and older (at least 12 months since last menstrual cycle)
* Participant in physical activity (e.g., 2-4 bouts of physical activity per week (i.e., activities such as brisk walking, yoga, hiking, cycling, gardening, etc.)) -Participants taking hormone replacement therapy (HRT; at least 6 months on HRT), statins, and antihypertensive medications will be allowed to participate.

Exclusion Criteria:

* Food allergies
* Dietary restrictions (e.g., vegan, vegetarian, lactose intolerance, etc.)
* Diet-related conditions that would prevent them from consuming a higher protein dietary intake (e.g., impaired liver function, kidney disease)
* Participants consuming more than 0.8 g protein/kg/body weight per day (determined by 24-hour dietary recall)
* Underweight (BMI < 18.5)
* Taking nutritional supplements
* Currently smoking or vaping
* Use marijuana
* Drink more than 4 alcoholic beverages a week
* Take medications that may interfere with the primary outcomes of the dietary intervention (e.g., antidepressants, sleep medication, etc.)
* Sleep apnea
* Pittsburgh Sleep Quality Index (PSQI) global score >5 via or sleep > 7 hours a night
* Pre-existing health conditions (e.g., diabetes (type I or II), cancer, Parkinson's Disease, Multiple Sclerosis) or conditions that would prevent them from fully participating in all aspects of the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality and Duration | 16 weeks
  Sleep quality and duration will be assessed objectively via an ActiGraph triaxial wrist accelerometer GT9X Link (ActiGraph, LLC, Pensacola, FL, USA), a validated method of sleep assessment. Each participant will wear an ActiGraph monitor on the non-dominant wrist for 24 hours/day for seven days (except when bathing or involved in water activities) prior to the start of the intervention and every four weeks throughout the intervention. Accelerometers will be fitted securely on each participant's wrist. Participants will receive sleep diaries to define "time in bed" and "time out of bed." The indicated "start" and "end" points will be used to define a sleep region to be analyzed within the ActiGraph software. Sleep outcomes will be calculated based on epoch-to-epoch sleep/wake algorithms within the defined sleep period. Data will be processed by using the ActiLife Version 6.9.2 software (Pensacola, FL, USA) and sleep will be scored via the Cole-Kripke algorithm. The following
Mood | 16 weeks
  The Profile of Mood States (POMS) questionnaire will be used to assess mood. POMS consists of 65 questions containing a one-word adjective of mood to measure and identify six affective states. The six identifiable mood/affective states are tension-anxiety, depression-dejection, anger-hostility, vigor-activity, fatigue/-inertia, and confusion-bewilderment. Participants will be instructed to define their mood on a 5-point Likert scale ranging from 0 to 4. The numbers refer to the following descriptive phrases: 0 = Not at all, 1 = A little, 2 = Moderately, 3 = Quite a bit, 4 = Extremely. Prior to the start of the questionnaire each participant will read the following directions: Describe how you have been feeling during the past week including today by circling the number that best describes your present mood with 0 indicating "Not at all," and 4 indicating "Extremely".
Qualify of Life Assessment | 16 weeks
  Quality of life assessment (QoL) will be measured using the SF-36 questionnaire. The SF-36 relies on participant self-reporting and measures 8 QOL domains which are dichotomized into physical (functioning, role limitations-physical, pain, general health) and mental health (vitality, social functioning, role limitations-emotional, and emotional/mental health). Item scores are converted to a 0-100-point scale; domain scores are derived by averaging individual items within the subscale; and physical composite and mental health composite scores were derived by averaging the four component domains of each. Higher values are indicative of better QoL.

SECONDARY OUTCOMES:
Height | 16 weeks
  Height will be measured to the nearest 0.01 cm using a standard stadiometer.
Dietary intake | 16 weeks
  Dietary intake will be measured using 3-day, weighed food records.
Fat mass | 16 weeks
  Fat mass will be measured using dual x-ray absorptiometry.
Plasma amino acids | 16 weeks.
  Plasma amino acid profiles will be measured in the fasted state.
Fat-free mass | 16 weeks
  Fat-free mass will be measured using dual x-ray absorptiometry.
Bone mineral density | 16 weeks
  Bone mineral density will be measured using dual x-ray absorptiometry.
Weight | 16 weeks
  Body weight will be measured to the nearest 0.05 kg using a calibrated scale in the fasted state.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Baum, Principal Investigator — University of Arkansas System Division of Agriculture
Locations (2):
- United States (2):
  - Don tyson Center for Agricultural Sciencers, Fayetteville, Arkansas
  - University of Arkansas, Fayetteville, Arkansas

IPD SHARING:
Plan to Share IPD: Undecided
We are planning on sharing IPD but need approval of the plan by the University.